CLINICAL TRIAL: NCT03887663
Title: The Chinese Parkinson's Disease Registry
Brief Title: Chinese PD Registry
Acronym: CPDR
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CPDR
Record Dates: First submitted 2018-12-02; First posted 2019-03-25 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
Keywords: Motor symptoms; Nonmotor symptoms; Chinese longitudinal cohort; Natural history
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extraction of DNA from peripheral blood of patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese Parkinson's disease Registry (CPDR) is to develop a database of patients with Parkinson's disease in China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among degenerative neurological diseases. PD is a complicated disease which consists of different subtypes. A certain type of parkinsonism has its unique clinical feature and genetic basis. Standards of classification and prognosis in different PD subtypes are still poorly understood. Investigators aim to establish a database of longitudinal recruited PD cohort ,and characterize the clinical feature, genetic basis, environmental factors and their interactions among different PD subtypes in China, identify natural history of a highly-presentative Chinese PD cohort and to discern major milestones in the disease process which indicates disease progression.

Data were collected at baseline, 12±1 months during the routine follow-up visits. Information about detailed disease history, level of education, significant chronic comorbidities, physical examination, medication history, family history, living habits and toxic exposure history, which include smoking, drinking tea, alcoholic consumption, drinking coffee, exposure to pesticide or occupational solvent, history of carbon monoxide poisoning and recurrent head trauma will be recorded at baseline. For each evaluation, the same questionnaires will be conducted. A standardized neurological assessment according to the recommendation of Consensus on the construction of clinical database of Parkinson's disease and movement disorders in China. The Unified Parkinson's Disease Rating Scale (UPDRS) part III is conducted for motor assessment, all the patients are evaluated in "OFF" state. The clinical stage of PD is assessed by Hoehn and Yahr scale (H-Y). The non-motor symptoms are evaluated by Non-motor Symptom Scale (NMSS), autonomic symptoms are evaluated by The Scale for outcomes in Parkinson disease for Autonomic Symptoms (SCOPA-AUT). Constipation was diagnosed by Functional Constipation Diagnostic Criteria Rome Ⅲ. The 39-item Parkinson's Disease Qestionnaire (PDQ-39) was used to assess the quality of life. Sleep quality was evaluated by Parkinson's Disease Sleep Scale (PDSS) and excessive daytime sleepiness by Epworth Sleepiness Scale (ESS). Probable rapid eye movement sleep behavior disorder (p-RBD) was diagnosed by rapid eye movement sleep behavior questionnaire-Hongkong (RBDQ-HK). Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire (CH-RLSq). Cognitive assessment was used the previously validated scale, Mini Mental State Examination (MMSE). Olfaction test was carried out by Hyposmia Rating Scale (HRS), a proportion of patients was also ascertained by Sniffin's Sticks. Depression was diagnosed by Hamilton Depression Scale (HAMD). Symptom of fatigue was measured by PD fatigue severity scale (PFS). Wearing-off was evaluated by WOQ-9 and freezing gait by new freezing gait questionnaire scores (NFOGQ). Dyskinesis was evaluated by Rush Dyskinesia Rating Scale. DNA samples extracted from peripheral blood and all the PD patients will be examed by Whole Exome Sequencing or Whole-genome sequencing. All the participants are scanned by structural MRI to exclude obvious intracranial lesions and other parkinsonism such as MSA, PSP and WD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD by UK Brain Bank Diagnostic Criteria and other standard criteria.

Exclusion Criteria:

* Lack of capacity to consent to participate in the project

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Most of the PD patients comes from mainland China, especially from Hunan Province, Hubei Province, Jiangxi Province and Guizhou Province. The proportion of male patients is slightly dominant than that of female patients. The age of PD patients ranges from 13 to more than 90 years old.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale for evaluating motor subtypes | 12±1 months
  The UPDRS is made up of four parts, 55 items in total. Total score varies from 0 to 199. Part I: evaluation of behavior and mood, which consists of 4 items, score varies from 0-16; Part II: self-evaluation of the activities of daily life, which consists of 13 items,score varies from 0-52; Part III: motor evaluation, which consists of 27 items, score varies from 0-108; Part IV: complications of therapy, which consists of 11 items,score varies from 0-23. All the patients are evaluated in "OFF" state. The ratio of the mean tremor score (scores of item-16, item-20, and item-21 will be added: ) to the mean postural instability/gait disorder (PIGD) score (scores of item-13, item-14, item-15, item-29, item-30 will be added: ) was used to classify motor subtype. Patients with a ratio value < 1.0 were defined as PIGD, and those with values from 1.0 to 1.5 were categorized as intermediate, while those with values ≥1.5 were classified as tremor dominant.
The clinical stage of PD is assessed by Hoehn and Yahr scale | 12±1 months
  The H-Y scale ranges from 1 to 5. Early PD is defined as H-Y stage 1 to 2.5, advanced PD is defined as H-Y stage 3-5.
Autonomic symptoms are evaluated by The Scale for outcomes in Parkinson disease for Autonomic Symptoms | 12±1 months
  This scale includes 25 items assessing the following regions: gastrointestinal (7 items), urinary (6 items), cardiovascular (3 items), thermoregulatory (4 items), pupillomotor (1 items), and sexual dysfunction(2 items for men and 2 items for women). Scores in each region should be added. The score of the answers ranges from 0 to 3 for each item and the total score ranges from 0 to 69, where higher scores reflect worse autonomic functioning.
The non-motor symptoms are evaluated by Non-motor Symptom Scale | 12±1 months
  This scale includes 30 items which is divided into 9 domains. Total score varies from 0-360. Higher score indicates severer symptoms. Domain 1 evaluates cardiovascular system symptoms. Score of domain 1 varies from 0-24. Domain 2 evaluates sleep condition. Score of domain 2 varies from 0-48. Domain 3 evaluates cognitive function. Score of domain 3 varies from 0-72. Domain 4 evaluates illusion. Score of domain 4 varies from 0-36. Domain 5 evaluates attention and memory. Score of domain 5 varies from 0-36. Domain 6 evaluates gastrointestinal symptoms. Score of domain 6 varies from 0-36. Domain 7 evaluates urinary symptoms. Score of domain 7 varies from 0-36. Domain 8 evaluate sensory symptoms. Score of domain 8 varies from 0-24. Domain 9 evaluates other non-motor symptoms. Score of domain 9 varies from 0-48.
Constipation was diagnosed by Functional Constipation Diagnostic Criteria Rome III. | 12±1 months
  The diagnostic criteria must include two or more of the following
  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools in at least 25% of defecations
  3. Sensation of incomplete evacuation for at least 25% of defecations
  4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
  5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
  6. Fewer than three defecations per week 2. Loose stools are rarely present without the use of laxatives 3. Insufficient criteria for irritable bowel syndrome * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
The PDQ-39 was used to assess the quality of life. | 12±1 months
  This scale includes 39 items assessing the following regions: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communications (3 items) and bodily discomfort (3 items). Alternatively, the sum of the scores can assess the overall health-related quality of life profile of the individual questioned. Scores in each region should be added. The score of the answers ranges from 0 to 4 for each item and the total score ranges from 0 to 116, where higher scores reflect worse life quality.
Sleep quality is evaluated by Parkinson's Disease Sleep Scale | 12±1 months
  This scale includes 15 items that address eight aspects of sleep disturbances in PD, including overall quality of night's sleep (item 1)), score of item 1 less than 6 is defined as sleep disorder. Score of all the questions will be summed. The score of the answers ranges from 0 to 10 for each item and the total score ranges from 0 to 150, where higher scores reflect better sleep condition.
Excessive sleepiness is evaluated by Epworth Sleepiness Scale | 12±1 months
  This scale includes 8 items. Score of all the questions will be summed. All items were rated on a 4-point scale (0-3), with a minimal score of 0, and maximum total score of 24. A higher score demonstrates more severe excessive daytime sleepiness. Participants were classified as showing excessive daytime sleepiness if their total score ≥10 .
Probable rapid eye movement sleep behavior disorder was diagnosed by Probable rapid eye movement sleep behavior disorder Questionnaire -Hongkong | 12±1 months
  This scale includes 13 items. Score of all the questions will be summed. Total score of the answers ranges from 0 to 100, where higher scores reflect severer rapid eye movement sleep behavior disorder.The optimal cutoff value for the overall scale is 17; subjects were classified as showing RBD when they reached the above score.
Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire | 12±1 months
  1. have, or have you had, recurrent uncomfortable feelings or sensations in your legs while you are sitting or lying down
  2. have, or have you had, a recurrent need or urge to move your legs while you were sitting or lying down
  3. more likely to have these feelings when you are resting
  4. If you get up or move around when you have these feelings, these feelings get better
  5. these feelings in your legs most likely to occur at mid-day or afternoon or evening or night
  6. Simply changing leg position by itself once without continuing to move usually relieve these feelings usually don't relieves
  7. These feelings are not or not always due to muscle cramps
Cognitive condition is assessed by Mini Mental State Examination | 12±1 months
  This scale includes 30 items. Score of all the questions will be summed. All items were rated on a 2-point scale (0-1), with a minimal score of 0, and maximum total score of 30. A higher score demonstrates more better cognitive condition. The definition of cognitive disorder differs in education level. For illiteracy, presence of cognitive impairment is defined as MMSE score. For those only receive elementary education, the cut-off value is 20. For other patients, presence of cognitive impairment was defined as MMSE scores less than 25.
Olfaction test was measured by Hyposmia Rating Scale | 12±1 months
  This scale includes 6 items. Score of all the questions will be summed. All items were rated on a 4-point scale (1-4), with a minimal score of 6, and maximum total score of 24. A higher score demonstrates more worse sense of olfaction. The cutoff value HRS is 22.5.
Depression was diagnosed by Hamilton and Montgomery-Asberg Depression Scale | 12±1 months
  This scale includes 17 items. Score of all the questions will be summed. Total score ranges from0-53. A higher score demonstrates more severer depression. The study participants were defined to be not depressed (scores 0-6) , to have minor depression(scores 7-14), or to have major depression (scores above 14) at the different visits during follow-up
Symptom of fatigue was measured by PD fatigue severity scale | 12±1 months
  This scale includes 9 items. Score of all the questions will be summed. All items were rated on a 7-point scale (1-7). Total score ranges from0-63. A higher score demonstrates more severer fatigue.
freezing gait by new freezing gait questionnaire scores | 12±1 months
  Parts II and III provides a total summed score between 0 and 28. Part II (items 2-6, scoring range 0-19) rated the severity of FOG based on its duration and frequency in its most common manifestation. Total score will be calculated for comparison.
Dyskinesia was evaluated by UPDRS part III | 12±1 months
  The presence of dyskinesia is evaluated by the doctor and recordsed.

SECONDARY OUTCOMES:
hypertension | baseline
  Diastolic blood pressure ≥140 mmHg, or systolic blood pressure ≥90 mmHg in at least three different days; or self-reported hypertension diagnosed by physicians, or taking BP-lowering medications at baseline.
Type II diabetes | baseline
  Type II diabetes can be diagnosed if any of the requirements are met: The test result of serum Hemoglobin A1c level conducted in the hospital is higher than 6.5%, fasting plasma glucose level ≥7.0mmol/l, or oral glucose tolerance test results ≥11.1mmol/l, results confirmed by repeated testing, or random plasma glucose level ≥11.1mmol/l in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis; or self-reported type II diabetes diagnosed by physicians, or taking hypoglycemic agent or insulin at baseline.
Hyperlipidemia | baseline
  Total cholesterol ≥6.2mmol/L or low-density lipoprotein ≥4.1mmol/L or triglyceride ≥2.3mmol/L; or self-reported hyperlipidemia diagnosed by physicians, or taking lipid-lowering drugs at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changzhi, Hunan, China